CLINICAL TRIAL: NCT01824108
Title: Effectiveness of Wallis Interspinous Dynamic Stability System for Lumbar Disc Herniation: a Prospective Randomised Controlled Study
Brief Title: Wallis Interspinous Dynamic Stability System for Lumbar Disc Herniation: a Prospective Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Qiujiang Zheng, Director of Orthopaedic Surgery, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WALLIS-2008
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar disc herniation; Wallis interspinous implants; lumbar discectomy; interspinous dynamic stability system
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group: Lumbar discectomy (Active Comparator): Lumbar discectomy alone
  Interventions: Procedure: Lumbar discectomy
- Treatment group: lumbar discectomy + Wallis implant (Experimental): lumbar discectomy combined with Wallis interspinous dynamic stability system
  Interventions: Procedure: Lumbar discectomy combined with Wallis interspinous dynamic stability system

INTERVENTIONS:
Procedure: Lumbar discectomy — All the patients were in prone positions on the operation table and received general anesthesia. A midline incision was made and paravertebral muscles were dissected unilaterally. Disc excision and nerve root decompression were initially accomplished through a unilateral transflaval approach. Then the wound was closed with a suction drain.
  Arms: control group: Lumbar discectomy
Procedure: Lumbar discectomy combined with Wallis interspinous dynamic stability system — The Wallis interspinous implant is placed after a lumbar discectomy. Interspinal ligaments of operated segment were removed and supraspinal ligament were retained. And then the proper size of Wallis implant was mounted underneath the supraspinous ligament and secured to the spine with the attached Dacron bands,above and below the corresponding spinous processes.
  Arms: Treatment group: lumbar discectomy + Wallis implant

SUMMARY:
Lumbar disc herniation is usually treated by discectomy alone. Nonfusion system such as Wallis interspinous implants have also been successfully used in disc degenerative diseases. However, the superiority of a discectomy with Wallis in comparison to a discectomy alone for primary lumbar disc herniation has yet to be determined.The aim of our study is to investigate whether lumbar discectomy combined with the Wallis device provides better radiographic and clinical short-term outcome than posterior lumbar discectomy alone.

DETAILED DESCRIPTION:
The most commonly used therapy for lumbar disc herniation (LDH) are partial discectomy or discectomy with fusion if there was an additional mechanical disorder in the underlying functional spinal unit. However, the problems associated with discectomy are intervertebral disc height loss and the segmental instability, thought to be a risk for failed back surgery syndrome or recurrence lumbar disc herniation. Fusion has also been criticised for its side effects of adjacent segment degeneration(ASD), pseudarthrosis and bone-graft morbidity. To prevent such complications , a new family of dynamic implants have been established. Wallis interspinous implant (Abbott Laboratories, Bordeaux, France) , invented by J. Senegas, is one of them. It consisted of a interspinous blocker made out of polyetheretherketone (PEEK) to limit extension and two dacron tapes around the spinous processes in order to secure the implant and limit flexion. The aim of using this device is to unload the facet joints, to restore foraminal height and to provide sufficient stability especially in extension but still allow motion in the treated segment. Previous clinical trials and biomechanical studies are promising, however, the superiority of a discectomy with Wallis in comparison to a discectomy alone for primary lumbar disc herniation has yet to be determined. The purpose of this prospective controlled study was to evaluate the clinical effect of lumbar discectomy combined with Wallis interspinous device, comparing with posterior lumbar discectomy alone. Our hypothesis was that the use of the Wallis device would have better clinical and radiological outcomes than lumbar discectomy alone.

ELIGIBILITY:
Inclusion criteria:

1. 18-70 years old;
2. complaining low back pain or radioactive melosalgia;
3. preoperative image examination showing disc herniation or spinal stenosis caused by herniation of responsible level;
4. no improvement in symptoms after 6-10 weeks of non-surgical treatment.

Exclusion criteria:

1. previous operations;
2. congenital spinal deformity;
3. lumbar fracture;
4. infection;
5. autoimmune diseases;
6. serious osteoporosis;
7. morbidly obese;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) at 2 days before intervention | 2 days before intervention
  baseline VAS
Visual Analogue Scale (VAS) at 1 week after intervention | 1 week after intervention
Visual Analogue Scale (VAS) at 12 months after intervention | 12 months after intervention
Visual Analogue Scale (VAS) at 24 months after intervention | 24 months after intervention
Japanese Orthopedics Association (JOA) at 2 days before intervention | 2 days before intervention
  baseline JOA
Japanese Orthopedics Association (JOA) at 1 week after intervention | 1 week after intervention
Japanese Orthopedics Association (JOA) at 12 months after intervention | 12 months after intervention
Japanese Orthopedics Association (JOA) at 24 months after intervention | 24 months after intervention
Oswestry Disability Index (ODI) at 2 days before intervention | 2 days before intervention
  baseline ODI
Oswestry Disability Index (ODI) at 1 week after intervention | 1 week after intervention
Oswestry Disability Index (ODI) at 12 months after intervention | 12 months after intervention
Oswestry Disability Index (ODI) at 24 months after intervention | 24 months after intervention

SECONDARY OUTCOMES:
Intervertebral disc height of the operated segments | 2 days before intervention and 1 week, 12 months and 24 months after intervention
Range of motion of the operated segments | 2 days before intervention, 12 months and 24 months after intervention
Complications | 1 week, 12 months and 24 months after intervention
  Complications: includes dural laceration, implant loose, lumbar kyphosis, spinous process fracture or recurrent lumbar disc herniation

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Gerneral Hospital, Guangzhou, Guangdong, China